Cover page with the Official Title of the study: An Internet-based Self-help Intervention for the Reduction of Consumption of Ultra-processed Products and Increase of Physical Activity in Mexican University Population: Study Protocol for a Randomized Controlled Trial. Date:

April 9th, 2023

### Informed consent

A group of researchers from the University of Twente, the University of Guadalajara (UDG), and collaborating institutions, are conducting a study with the aim of implementing a self-applied online intervention based on scientific evidence for the acquisition of knowledge in the adoption of a healthy diet and physical activity to counteract the impact on psychopathological symptoms derived from the contingency by COVID-19.

Before you decide whether or not to participate, you should know and understand each of the following sections. This process is known as informed consent. Feel free to ask about any aspect that helps you clarify your doubts about it. Once you have understood the study and if you want to participate, you will then be asked to click accept consent.

## Rationale for the study

One of the main effects on the university population after the covid-19 pandemic has been the changes in diet. This intervention is aimed at the Mexican university population that was in confinement due to the COVID-19 pandemic.

# **Objective of the intervention**

That the participant acquires knowledge in the adoption of a healthy diet and physical activity to counteract the impact on psychopathological symptoms derived from the COVID-19 contingency.

### **Procedure**

The intervention is composed of 9 interconnected modules and 2 follow-up modules, one for 3 months and the last one for 6 months, to which you will have access when registering on the platform. To register on the platform, it is only necessary to provide your email. At no time during the study will you be asked for other types of information or sensitive or personally identifiable data such as your name, telephone number, address.

Prior to the start of the modules, you will be asked to carry out a brief evaluation which consists of a series of questions, as well as various psychometric instruments that will take 30-35 minutes. If there is a question that you do not understand, please notify the responsible investigator by email and continue with the next question. The important thing is that you answer exactly what is happening in your case, because that is precisely what we want to know. There are no right or wrong questions, so please answer as honestly as possible.

After the assessment, you will be able to access each of the modules that constitute the intervention.

#### **Risks**

In accordance with the Regulations of the General Health Law on Health Research, this intervention is considered to have minimal risk, this means that only some psychological tests will be applied in which the subject's behavior will not be manipulated. not having affectation in the participating subjects..

## Willfulness

Your participation in this study is completely voluntary, so you are free to stop participating in the study at any time. This program is totally free being part of the benefits of the study. And to be able to carry it out, we only ask you to have an internet connection and a device so that you can connect regularly and be able to carry out the intervention modules.

# Confidentiality

The results of this research will be analyzed for research purposes and, therefore, may be published in scientific journals, books or disseminated by other means to the scientific community, taking care at all times of the confidentiality and anonymity of the data of the participants. This study has the approval of the research ethics committee of the University of Guadalajara of the University Center of Health Sciences.

All information generated will be treated confidentially. Your identification data will not appear in the databases since only a participant page will be shown. In the final report of the study, in the publication of results in scientific congresses, in publications in scientific journals and at all times, your identity will remain anonymous. To guarantee the confidentiality and protection of your personal data, all forms and questionnaires will only have one code randomly assigned and they will not contain any type of personal data that could serve to identify you, not even by date of participation, adress, etc.

# Benefits that you will obtain by participating

If you accept your participation, you will receive a self-applied online intervention, based on scientific evidence and completely free at all times, through a program of 9 interactive modules and 2 follow-up ones.

If you agree with the above, we invite you to click accept. If you do not participate, you can close your internet window.

In this application, you inform that you agree to voluntarily participate in this research that we are conducting and, therefore, are willing to complete the questionnaires. In addition to the above, it is important to clarify that:

- I can request information about the study at any time during the process.
- I can contact the people who are applying this series of questionnaires to dispel my doubts regarding the research.

I understand that my participation is voluntary and that I can withdraw from the study:

- Whenever I want
- Without having to explain
- Without this affecting my integrity as a person
- I freely give my consent to participate in the study.

If you have any questions, doubts, comments or concerns regarding the intervention, please contact fabiola.macias@academicos.udg.mx, principal investigator, where we guarantee to receive a response to whatever your concern may be.

I freely give my consent to participate in the study:

yes I agree to participate

I do not accept to participate

Please select the appropriate option or complete the space with the following information, as the case may be.